CLINICAL TRIAL: NCT05796466
Title: Improving Vulnerable Preschoolers' Mental Health: A Superiority Trial Assessing the How-to Parenting Program
Brief Title: Improving Preschoolers' Mental Health: A RCT Assessing Two Parenting Programs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mireille Joussemet (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Mireille Joussemet, Associate Professor, Université de Montréal
Organization: Université de Montréal (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: How-to_preschool
Record Dates: First submitted 2023-03-04; First posted 2023-04-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Mental Health Issue; Parenting
Keywords: Parenting program

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will only know the name of the parenting program they are taking part of, but the name of the other program will not be disclosed. All research assistants who will conduct evaluations (i.e., observational tasks) or code parent-child interactions will be blind to experimental assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- How-to Parenting Program (Experimental): The How-to Parenting Program is a highly structured and skill-based program. It is manualized, teaches 30 concrete, specific, easy-to-grasp (e.g., taught using comic strips), and readily applicable skills. It also optimizes learning with exercises (e.g., perspective taking; role-playing) and practice, and addresses parents' readiness and motivation to change. The program is delivered over six consecutive 2-hour weekly sessions (12 hours in total).
  Interventions: Behavioral: How-to talk so kids will listen and listen so kids will talk
- Nobody's Perfect Program (Active Comparator): Based on andragogy principles, parents following the Nobody's Perfect curriculum will learn how to solve problems with their child and engage in theme-related activities meant to increase awareness of parents' own needs, child behaviors, development, health, and safety. There is no pre-determined order for themes and time devoted to each one varies according to parents' needs. The program is delivered over six consecutive 2-hour weekly sessions (12 hours in total).
  Interventions: Behavioral: Nobody's Perfect

INTERVENTIONS:
Behavioral: How-to talk so kids will listen and listen so kids will talk — The How-to Parenting Program focuses on how expectations, rules, and values are better communicated (vs. what rules ought to be). It includes skills related to the three components of authoritative parenting, namely affiliation, structure, and autonomy support. 1) Affiliation: Parents learn how to listen and respond to their children in a way that helps them feel accepted unconditionally. 2) Structure: Parents learn how to communicate expectations, give feedback, follow through, and use joint problem-solving in a factual, non-judgmental way. 3) Autonomy support: Parents learn how to validate emotions, encourage initiatives, and free children from roles. Finally, the How-to program can be endorsed by parents of various cultural backgrounds, as suggested by the large number (> 30) of languages in which the material is translated. This advantage is crucial in ethnically diverse regions such as Canada.
  Other Names: How-to Parenting Program
  Arms: How-to Parenting Program
Behavioral: Nobody's Perfect — Nobody's Perfect is delivered in family resource centers across Canada to support parents of infants and preschoolers. Its focus is on developing parents' capacity to problem solve, providing child development information, and helping parents recognize their strengths and find their own positive ways to interact with their children. It thus does not teach specific parenting skills and does not suggest specific rules to put into practice in the home-environment.
  Arms: Nobody's Perfect Program

SUMMARY:
The goal of this randomized control trial (RCT) is to assess the superiority of the How-to Parenting Program in improving autonomy support and preschoolers' mental health (i.e., decreases externalizing problems) among vulnerable families. The main question it aims to answer is: Can teaching concrete parenting skills that target empirically-based parenting dimensions (via the How-to Parenting Program) have an added value for improving parental autonomy support and child mental health, compared to a parenting program that does not focus on teaching parenting skills (Nobody's Perfect program [NP])? Early childhood centers providing services to parents of 3-4 years olds will be randomly assigned to one of two 6-week programs. Parents will fill out questionnaires before (T1) and after (T2) programs delivery as well as at 6-month (T3) and 1-year follow-ups (T4). They and their child will also engage in filmed parent-child interactions at T1 and T3 during predetermined activities, to obtain observational measures of parenting and child socioemotional competences. Researchers will compare the How-to and NP conditions to see if there was an accentuated increase in parental autonomy support and child mental health in the How-to condition. As secondary analyses, researchers will compare the How-to and NP conditions on parenting quality, child socioemotional competences, and parental cognitions as well as explore the conditions in which NP could be equal (or superior) to the How-to Parenting Program.

DETAILED DESCRIPTION:
This RCT with a 1-year follow-up aims to assess the superiority of the How-to Parenting Program in improving parental autonomy support and preschoolers' mental health (i.e., decreases externalizing problems) among vulnerable families. One out of five children younger than age 7 presents mental disorders. Without proper help, such difficulties impede later health and functioning, making early intervention aimed to reduce mental health problems a social imperative.

Among environmental factors, parenting quality is the most widely accepted predictor of child mental health. Decades of parenting research show that parenting quality has three components fostering child development and mental health: affiliation, structure, and autonomy support. Investigators aim to assess the impact of the How-to Parenting Program, an accessible program that addresses all components of parenting quality. Reseacrhers will compare it to the Nobody's Perfect (NP) program, a program delivered in communities across Canada that is similar in format (6 weekly group sessions), similar in cost (no costly certification), but different in content (NP does not focus on parenting skills).

In a prior wait-list RCT with school-aged children, investigators found that the How-to Parenting Program improved both parenting quality and child mental health. The present RCT aims to test whether teaching concrete parenting skills that target empirically-based parenting dimensions (via the How-to Parenting Program) improves parental autonomy support and the mental health of younger children to a greater extent than the NP Program.

Investigators will recruit 320 parents of 3- and 4-year-olds from a large pool of early childhood centers (ECCs; i.e., family resource centers and daycares). At each of five yearly waves, ECCs will be randomized to the experimental condition (4 How-to groups; ≈ 32 parents) or the active control condition (4 NP groups; ≈ 32 parents). Parents will fill out questionnaires before (T1) and after programs delivery (T2) and at 6-month (T3) and 1-year follow-ups (T4). Both programs will be delivered online, by two trained facilitators. Parents, blind to their condition allocation, will rate their child's mental health problems and their autonomy-supportive behaviors (primary outcomes) as well as their child's socio-emotional competencies, and other parental behaviors and cognitions. Parent-child filmed interactions will allow observational measures of child self-regulated behaviors and parenting quality). Based on prior findings, investigators expect greater improvements in parental autonomy support and child mental health in the How-to condition compared to the NP condition. Investigators also expect larger improvements on secondary outcomes in the How-to condition, with the exception of the parental cognitions specifically targeted by NP (problem-solving; social support). Finally, researchers expect both programs to have similar benefits for among more vulnerable parents.

By evaluating the added benefits of the How-to Parenting Program, this research will reduce the know-do gap, helping practitioners and other stakeholders to make evidence-based decisions regarding the delivery of helpful parenting interventions to improve preschoolers' mental health.

ELIGIBILITY:
Inclusion Criteria:

- Parents need to have at least one child aged between between 36 and 59 months at pre-intervention.

Exclusion Criteria:

* Parents will be excluded if they have previously attended a How-to Parenting Program
* Parents who are unable to communicate in French will be excluded.

Recruitment procedure:

- To target more more vulnerable families, parents will primarily be recruited in ECCs located in low- or middle-income neighbourhoods of the greater Montreal (Canada) according to the Montreal's 2018 Poverty Map of Families with Children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2029-06-15 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in children's externalizing problems | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will complete the externalizing scale of the Child Behavior Checklist (Achenbach et al. 2001) for ages 1.5 to 5. The scale is answered on a 3-anchor rating scale ranging from "does not apply (as far as you know)" to "always or often applies". The externalizing scale comprises 24 items on aggressive and attention problems.
Change in parental autonomy support | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will answer seven items of the Parental Attitude Scale (Grolnick et al., 1997) to rate their attitude toward autonomy support and controlling parenting. This scale has predictive validity and has been associated with observational measures of autonomy-supportive and controlling behaviors. The scale is answered on a 7-anchor Likert scale ranging from "do not agree at all" to "very strongly agree".

SECONDARY OUTCOMES:
Change in observed parenting practices | Baseline and 8-month follow-up.
  Parents' verbal and non-verbal behaviors will be coded using a time-sampling coding scheme with mutually exclusive categories. To control for parents' propensity toward social interactions, each parenting component will be examined in relation to the number of coded behaviors.
  A total of 50 behaviors will be coded (Labelle et al., 2023), selected based on previous coding systems (Eisenberg et al., 2010; Robinson & Eyberg, 1981; Laurin & Joussemet, 2017) and past literature (e.g., Reeve, 2009).
  Affiliation: Parental sensitive availability/warmth.
  Rejection: Cold and rejecting behaviors.
  Structure: Feedback (Confirming), non-solicited guidance (Non-solicited questions) & solicited guidance (Solicited information or hints).
  Chaos: Incompetent/chaotic guidance (Misleading guidance)
  Autonomy support: Empathic behaviors & choice (Following child's initiative).
  Controlling behaviors: Task-related (Directives) & psychological control (Task-related criticisms; Orders).
Change in observed child committed compliance | Baseline and 8-month follow-up.
  We will use Kochanska's coding scheme to code committed compliance (eagerly or spontaneously pick up toys, beams or claps hands after putting toys in the box), situational compliance (halfheartedly cooperates after being prompted, attention shifts back to playing), and defiance (ignores parental prompts, negotiations, resistance, and oppositional behaviors).
Change in children's socio-emotional competencies | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will fill the Devereux Early Childhood Assessment (DECA; LeBuffe & Naglieri, 1999). The DECA is a standardized, norm-referenced, behavior rating scale for ages 2 to 5. It evaluates child social and emotional competences (initiative, self-control, and trust) with 26 items. Parents are asked to respond on a 7-point rating scale (ranging from "almost never" to "almost always") how often their child exhibits specific behaviors.
Change in children's internalizing problems | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will complete three of the internalizing subscales of the Child Behavior Checklist (Achenbach et al. 2001) for ages 1.5 to 5. Items are answered on a 3-anchor rating scale ranging from "does not apply (as far as you know)" to "always or often applies". The global internalizing score will comprise 25 items, the 3 subscales are anxious/depressed, emotionally reactive, and withdrawn.
Change in parental self-compassion | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will report their levels of self-compassion with the short version of the Self-Compassion Scale (Raes et al., 2011), which includes 12 items. The items are answered on a 7-anchor scale ranging from "almost never " to "almost always".
Change in parental efficacy | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will complete the efficacy subscale of the Parenting Sense of Competence scale (PSOC). Parents indicate their level of agreement with each item (e.g. I honestly believe I have all the skills necessary to be a good mother/father to my child) by rating a 7-anchor Likert scale ranging from "do not agree at all" and "very strongly agree".
Change in parental guilt | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will answer a questionnaire assessing their parental guilt by filling an Expanded Form of the Positive and Negative Affect Schedule (PANAS-X) Guilt subscale (Watson & Clark, 1991, 1994). The questionnaire includes 6 items and is answered on a 5-anchor scale ranging from "very little or not at all" to "extremely".
Change in parental stress | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will report the extent to which they experience stress in their daily lives using 4 items of the Perceived Stress Scale (e.g. Have you felt difficulties were piling up so high that you could not overcome them?") by rating a 7-anchor scale ranging from "almost never " to "almost always".
Change in parental social support | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will answer 4 questions of the Social Provisions Scale (Cutrona & Russell, 1987) to assess their perceived social support. The items are answered on a 7-anchor Likert scale ranging from "do not agree at all" to "very strongly agree".
Change in parental problem solving strategies | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will answer 4 questions on the Social Problem-Solving Scale (D'Zurilla, et al., 2002) to assess their problem solving strategies with their child. The items are answered on a 7-anchor scale ranging from "almost never" to "almost always".

OTHER OUTCOMES:
Change in parental perspective taking | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will complete 4 items of the perspective-taking subscale of the Interpersonal Reactivity Index (Davis, 1980), adapted to the mother-child relationship. Parents indicate their level of agreement with each item (e.g. Before criticizing my child, I try to imagine how I would feel if I were in his/her place) by rating a a 7-anchor Likert scale ranging from "do not agree at all" and "very strongly agree".
Change in parental emotional regulation | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will report the extent to which their emotional regulation strategies using the short version of the Emotional Regulation Scales (Roth et al., 2009). Three 4-item subscales assess dysregulation (e.g., When I feel negative emotions, I show them even in situations that are not appropriate for it.), suppressive regulation (e.g., I try to ignore negative emotions.), and integrative regulation (e.g., On occasions, negative emotions helped me to understand something about the situation I was in. The scale is answered on a 7-anchor Likert scale ranging from "do not agree at all " to "very strongly agree".
Change in parental social cohesion | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will report on the social cohesion they feel in their neighbourhood using 4 items (e.g., I borrow things and exchange favors with my neighbours) of the the Neighborhood Cohesion Instrument (Buckner, 1988). The scale is answered on a 7-anchor Likert scale ranging from "do not agree at all " to "very strongly agree".
Change in autonomy-supportive practices | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will report their tendency to adopt different autonomy-supportive behaviors with their child, using 10 items (e.g., When I ask my child to do something he/she doesn't like doing [e.g., getting dressed, taking a bath, picking up the toys], I offer to choose between two different ways of doing it) proposed by Andreadakis and her colleagues (2018). The scale is answered on a 7-anchor Likert scale ranging from "do not agree at all " to "very strongly agree".
Change in parental affiliation | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will answer 10 items of the Parental Bonding Instrument (Parker et al., 1979). The items are answered on a 7-anchor Likert scale ranging from "do not agree at all" to "very strongly agree".
Change in parental structure | Baseline, 2-month follow-up, 8-month follow-up, and 14-moth follow-up.
  Parents will answer four items (one per subscale) of the Multidimensional Parental Structure Scale (Ratelle et al., 2016) and three items (reversed) of the chaos subscale of the Parents as Social Context Questionnaire (Skinner et al., 2005). The items are answered on a 7-anchor Likert scale ranging from "do not agree at all" to "very strongly agree".

CONTACTS AND LOCATIONS:
Overall Officials: Joussemet Mireille, Ph.D., Principal Investigator — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data is not planned to be openly available, yet the study is open to collaboration and shared initiatives.

REFERENCES:
- [Background] Joussemet M, Mageau GA, Larose MP, Briand M, Vitaro F. How to talk so kids will listen & listen so kids will talk: a randomized controlled trial evaluating the efficacy of the how-to parenting program on children's mental health compared to a wait-list control group. BMC Pediatr. 2018 Aug 2;18(1):257. doi: 10.1186/s12887-018-1227-3. PMID 30071843
- See also: Protocol of a waitlist RCT assessing the How-to Parenting Program on school-aged children and their parents — https://doi.org/10.1016/j.appdev.2021.101383